CLINICAL TRIAL: NCT05270291
Title: Infectious Etiology of Vomiting in Children With Presumed Acute Gastroenteritis in the Absence of Diarrhea
Brief Title: Infectious Etiology of Vomiting in Children With Presumed Acute Gastroenteritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Hanna Szajewska, Profesor, Medical University of Warsaw
Other Study IDs: Isolated vomiting etiology
Record Dates: First submitted 2022-02-18; First posted 2022-03-08 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Acute Gastroenteritis; Vomiting
Keywords: acute gastroenteritis; children; vomiting; enteropathogens
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: rectal swab — rectal swab

SUMMARY:
In children with acute gastroenteritis (AGE), vomiting often precedes diarrhea. To establish the diagnosis of AGE, enteropathogen detection typically relies on diarrheal stool samples. However, testing requires sufficient stool sample, which may not be easily available. Recent studies suggest that in children presenting to emergency departments with presumed AGE with isolated vomiting, an enteropathogen can be identified using rectal swabs and molecular diagnostic tests. The rate of enteropathogen detection in children with isolated vomiting due to AGE may differ in various populations. Using rectal swabs and molecular diagnostic tests, we plan to assess the proportion of children with isolated vomiting with presumed AGE in whom an enteropathogen can be identified.

This will be a prospective cohort study. Children younger than 5 years with presence of ≥3 episodes of vomiting due to presumed AGE, lasting no longer than 7 days before enrolment, will be recruited. A total of 198 participants will be recruited and a rectal swab will be collected. The participants will be contacted 14 days after enrollment to complete a survey regarding symptoms experienced during that period and to identify any additional clinical care.

ELIGIBILITY:
Inclusion Criteria:

* age 0-5-year-old
* presence of ≥3 episodes of vomiting due to presumed AGE at inclusion
* <7 days of symptoms at the time of inclusion
* signed written informed consent

Exclusion Criteria:

* anticipated inability to complete 14 days follow-up
* history of neutropenia (as rectal swabs are contraindicated)
* critically ill status requiring urgent medical intervention
* inability to provide a rectal swab for testing
* chronic gastrointestinal tract disorders such as inflammatory bowel disease, cystic fibrosis, coeliac disease
* immunodeficiency

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children younger than 5 years with presence of ≥3 episodes of vomiting due to presumed AGE, lasting no longer than 7 days before enrolment, will be recruited.
Sampling Method: Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of children with isolated vomiting with presumed AGE in whom an enteropathogen can be identified. | immediately after the procedure

SECONDARY OUTCOMES:
Types of pathogens detected based on presenting symptoms | immediately after the procedure
The proportion of children with isolated vomiting with alternative diagnosis | immediately after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cepinska A, Kolodziej M, Podsiadly E, Szajewska H. Infectious Etiology of Vomiting in Children With Presumed Acute Gastroenteritis in the Absence of Diarrhea: Protocol for a Cohort Study. JPGN Rep. 2022 Oct 25;3(4):e268. doi: 10.1097/PG9.0000000000000268. eCollection 2022 Nov. PMID 37168472